CLINICAL TRIAL: NCT06708988
Title: Predictors of Outcome of Pediatric Renal Transplantation
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Merna Nazeer,MD, Assisstant Lecturer, Assiut University
Other Study IDs: Kidney transplantation
Record Dates: First submitted 2024-06-30; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Pediatric Renal Transplantation Complication
Keywords: pediatric renal transplantation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Renal transplantation is a unique chance to a normal life for end-stage renal disease patients, because of the perfect morphological and functional replacement of the lost kidneys. Serum creatinine and proteinuria reflect kidney allograft function, but they are nonspecific tools.Imaging techniques plays an important role in the detection of anatomical as well as functional abnormalities in the early stages.

DETAILED DESCRIPTION:
Renal transplantation is a unique chance to a normal life for end-stage renal disease patients, because of the perfect morphological and functional replacement of the lost kidneys. It is also the only effective way of replacement of the endocrine function of the kidneys. The survival of kidney grafts has improved considerably in recent years, due to advances in surgical techniques and in immunosupression protocols . Although improvements in surgical techniques and immunosuppression have led to longer survival, complications remain common, occurring in approximately 12%-20% of patients. Post transplantation complications can also be divided following the renal transplant's time of evolution into early complications (acute tubular necrosis, acute rejection, arterial or venous thrombosis, obstruction, urinary leak, post transplantation collections and infection) and late complications (transplant artery stenosis, arteriovenous fistulas, drugs toxicity, chronic rejection and urinary tract infection). Acute rejection (AR) is a major risk factor for chronic nephropathy and graft loss after renal transplantation (RT) . Antibody-mediated rejection (AMR) is the most common cause of allograft failure in kidney transplant recipients (KTRs) . Serum creatinine and proteinuria reflect kidney allograft function, but they are nonspecific tools. Despite its limitations (being invasive procedure with increased risk of bleeding and infection), kidney graft biopsy remains the gold standard method for confirming antibody-mediated rejection . Whilst kidney graft dysfunction could present with an elevated serum creatinine level, oliguria or pain over the graft site, it could also be asymptomatic. Imaging techniques plays an important role in the detection of anatomical as well as functional abnormalities in the early stages, thus allowing the chance for early treatment, as well as in the late post transplant period . Post-transplant complications can be divided into categories following the imaging-based classification of renal transplant complications: Perinephric collections, parenchymal abnormalities, abnormalities of the collecting system and vascular complications . The use of ultrasound to assess morphologic changes allows for the accurate and early detection of early pathologic alterations that may lead to rejection . Correlation of the ultrasound pattern with patient's history and clinical background is essential for a correct characterization. However, there are several limitations to ultrasound including its inability to assess renal function or differentiate between the different causes of renal dysfunction . Color Doppler ultrasonography, on the other hand, gives valuable information on the hemodynamics of the grafts' renal arteries. In the early post-transplant period, the resistive index(RI) measured in intrarenal arteries is thought to predict poor kidney graft performance . Doppler indices in different arteries differ in the detection of early parenchymal renal transplant complications. Resistive index of the interlobar artery proved to be more specific in the detection of early cases of parenchymal complications in a renal transplant patient . Color Doppler sonography had a limited value in the differentiation among the various etiologies of renal transplant dysfunction however the mean RI values were above normal in acute rejection and ATN . Vitamin D deficiency or vitamin D insufficiency is common and conflicting results concerning vitamin D deficiency -associated graft failure and mortality were described in kidney transplant recipients (KTRs). Many studies showed that Vitamin D deficiency , measured as 25-hydroxyvitamin D [25(OH)D] or 1,25-dihydroxyvitamin D [1,25(OH)2D], relates to kidney dysfunction in renal disease and graft loss in kidney transplant recipients . The association between low 1,25(OH)2D and graft failure was seen and was dependent on renal function. This association is not unexpected since the 1a-hydroxylase of the kidney, i.e., the enzyme that converts 25(OH)D into 1,25(OH)2D, is damaged simultaneously with the deterioration of renal function.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients aged 1 to 18 years old
* first renal transplant during the first year, pre and post complications.

Exclusion Criteria:

* patients with recurrent renal transplantation.
* Parental refusal to participate.
* Patients with chronic rejection

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All pediatric renal transplant recipients in their first year of transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
-Evaluation of pediatric renal patients during their first year after renal transplantation with doppler ultrasound by assessment of resistive index for early predictions of acute parenchymal rejection. | one year
-Evaluation of pediatric renal patients during their first year after renal transplantation with doppler ultrasound for early detection of vascular complications. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Maher Mokhtar, Professor, Study Director — Assiut University; Ahlam badwy, A.Professor, Study Director — Assiut University; Asmaa Ahmed, Lecturer, Study Director — Assiut University; Merna Ezzat, A. lecturer, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lim WH, Johnson DW, Teixeira-Pinto A, Wong G. Association Between Duration of Delayed Graft Function, Acute Rejection, and Allograft Outcome After Deceased Donor Kidney Transplantation. Transplantation. 2019 Feb;103(2):412-419. doi: 10.1097/TP.0000000000002275. PMID 29762458
- [Background] Takimoto Y, Imanaka F. [Chronic myelomonocytic leukemia with repeated respiratory failure associated with leukocytosis following splenic arterial embolization and splenectomy]. Rinsho Ketsueki. 1996 Nov;37(11):1253-8. Japanese. PMID 8960657
- [Background] Kim N, Juarez R, Levy AD. Imaging non-vascular complications of renal transplantation. Abdom Radiol (NY). 2018 Oct;43(10):2555-2563. doi: 10.1007/s00261-018-1566-4. PMID 29550956
- [Background] Bouatou Y, Viglietti D, Pievani D, Louis K, Duong Van Huyen JP, Rabant M, Aubert O, Taupin JL, Glotz D, Legendre C, Loupy A, Lefaucheur C. Response to treatment and long-term outcomes in kidney transplant recipients with acute T cell-mediated rejection. Am J Transplant. 2019 Jul;19(7):1972-1988. doi: 10.1111/ajt.15299. Epub 2019 Mar 15. PMID 30748089
- [Background] Schinstock CA, Mannon RB, Budde K, Chong AS, Haas M, Knechtle S, Lefaucheur C, Montgomery RA, Nickerson P, Tullius SG, Ahn C, Askar M, Crespo M, Chadban SJ, Feng S, Jordan SC, Man K, Mengel M, Morris RE, O'Doherty I, Ozdemir BH, Seron D, Tambur AR, Tanabe K, Taupin JL, O'Connell PJ. Recommended Treatment for Antibody-mediated Rejection After Kidney Transplantation: The 2019 Expert Consensus From the Transplantion Society Working Group. Transplantation. 2020 May;104(5):911-922. doi: 10.1097/TP.0000000000003095. PMID 31895348
- [Background] Mirzakhani M, Shahbazi M, Akbari R, Dedinska I, Nemati E, Mohammadnia-Afrouzi M. Soluble CD30, the Immune Response, and Acute Rejection in Human Kidney Transplantation: A Systematic Review and Meta-Analysis. Front Immunol. 2020 Feb 28;11:295. doi: 10.3389/fimmu.2020.00295. eCollection 2020. PMID 32256486
- [Background] Madubueze AG. Early Sonographic Evaluation of Intrarenal Arterial Resistive Index and Long-term Renal Function in Renal Transplant Recipients in South Western Nigeria. J Med Ultrasound. 2020 Mar 5;28(3):156-161. doi: 10.4103/JMU.JMU_82_19. eCollection 2020 Jul-Sep. PMID 33282659
- [Background] Galgano SJ, Lockhart ME, Fananapazir G, Sanyal R. Optimizing renal transplant Doppler ultrasound. Abdom Radiol (NY). 2018 Oct;43(10):2564-2573. doi: 10.1007/s00261-018-1731-9. PMID 30121777
- [Background] Meier M, Fricke L, Eikenbusch K, Smith E, Kramer J, Lehnert H, Nitschke M. The Serial Duplex Index Improves Differential Diagnosis of Acute Renal Transplant Dysfunction. J Ultrasound Med. 2017 Aug;36(8):1607-1615. doi: 10.7863/ultra.16.07032. Epub 2017 Apr 3. PMID 28370148
- [Background] de Braganca AC, Canale D, Goncalves JG, Shimizu MHM, Seguro AC, Volpini RA. Vitamin D Deficiency Aggravates the Renal Features of Moderate Chronic Kidney Disease in 5/6 Nephrectomized Rats. Front Med (Lausanne). 2018 Oct 10;5:282. doi: 10.3389/fmed.2018.00282. eCollection 2018. PMID 30370270
- [Background] Russell SE. Passing the hot potato--voluntary disclosure and Operation Restore Trust. Caring. 1996 Feb;15(2):36-9. No abstract available. PMID 10156982
- See also: Complications of renal transplantation: Diagnosis and treatment — https://dx.doi.org/10.1594/ecr2017/C-1274
- See also: ROLE OF RENAL ULTRASONOGRAPHY AND DOPPLER IN DETECTION OF COMPLICATIONS OF POST-TRANSPLANTED KIDNEY — https://dx.doi.org/10.21608/amj.2023.326112